

Document No. CL-003 Version 2.2 

# WISE LE Study protocol synopsis dated July 20 2016 NCT02780349

| Title: | WISE LE: Evaluation of WIRION™ EPS in Lower Extremities Arteries |
|---|---|
| Study Objective | Demonstrate the safety and performance of the WIRION™ EPS in subjects |
| | undergoing lower extremity atherectomy for the treatment of Peripheral |
| | Arterial Disease (PAD). |
| Study Design | Prospective, multi-center, non-randomized, open label, single arm study. Up to 153 consented subjects who undergo atherectomy due to lower limb PAD |
| | will be enrolled. All subjects will undergo baseline assessment, intervention |
| | (atherectomy in conjunction with WIRION <sup>TM</sup> EPS) and post procedure follow |
| | up. All subjects will have a follow up visit at 30±7 days post procedure. |
| | Results will be compared to a performance goal based on an analysis of |
| | previous trials that studied atherectomy with an embolic protection filter in |
| | similar patient cohorts. |
| Study Population: | Both male and female subjects who meet all the eligibility criteria and give written informed consent will be enrolled in the study. |
| | Inclusion Criteria |
| | 1) Subject is at least 18 years of age |
| | 2) Subject or authorized representative, signed a written Informed |
| | Consent form to participate in the study, prior to any study related |
| | procedures |
| | 3) Subject is willing to comply with the protocol requirements and |
| | return to the treatment center for all required clinical evaluations 4) Rutherford classification 2-4 |
| | 5) Has moderate to severe calcification visualized on angiogram in |
| | the femoropopliteal arteries |
| | 6) Planned atherectomy of the native femoropopliteal arteries |
| | 7) Reference vessel diameter for intended filter location must be |
| | visually estimated to be ≥3.5mm and ≤6.0mm |
| | 8) An adequate "landing zone" for placement of the WIRION™ device distal to the target lesion of at least 30mm |
| | 9) A female subject is eligible if not of child bearing potential or has a |
| | negative pregnancy test within the previous 7 days and agrees to |
| | remain on birth control throughout the study |
| | Exclusion Criteria |
| | <ol> <li>Any planned surgical or endovascular intervention within 30 days<br/>before or after the index procedure</li> </ol> |
| | 2) A lesion deemed not accessible by the WIRION™ EPS |
| | 3) Inability to take aspirin or ADP receptor antagonists |
| | 4) History of bleeding diathesis or coagulopathy or will refuse blood |
| | transfusion if deemed necessary |



Document No. CL-003 Version 2.2 

| Number of | <ul> <li>5) Has perforation, dissection, or other injury of the access or target vessel requiring additional stenting or surgical intervention before enrollment</li> <li>6) Subject is enrolled in another drug or device study protocol that has not reached its primary endpoint (participating in registry studies is not excluded)</li> <li>7) Life expectancy less than 12 months</li> <li>8) Known severe renal insufficiency (eGFR &lt;30 ml/min/1.72m²).</li> <li>9) ≤1-vessel tibial run-off status</li> </ul> |
|---|---|
| subjects: | Up to 153 with an interim analysis after 100 subjects |
| Clinical sites: | Up to 10 sites; up to 1/3 of the study patients at OUS sites |
| Investigational Product: | WIRION™ Embolic Protection System (Gardia Medical Ltd.) |
| | Freedom from major adverse events (MAE) to 30 days post procedure. |
| Primary end point | MAE defined as a serious adverse event that results in death, acute myocardial infarction, thrombosis, pseudo-aneurysm, dissection (grade C or greater) or clinical perforation at the filter location, distal embolism (clinically relevant), unplanned amputation, or clinically-driven target vessel revascularization (TVR), through 30 days post-procedure, as adjudicated by the Clinical Events Committee (CEC). |
| Secondary end points | <ul> <li>Device success Defined as: <ul> <li>A successful delivery and deployment of WIRION™ distal to the intervention site without complications, AND</li> <li>Successful retrieval of WIRION™ following completion of the stenting procedure, without complications</li> <li>Clinical success</li> <li>Defined as: Device success with freedom from procedure related serious adverse events ascribed to the WIRION</li> <li>Technical success</li> <li>Defined as: Freedom from device malfunctioning causing the procedure to be aborted</li> <li>Percent of filters with visible debris</li> </ul> </li> </ul> |
| Assessment<br>Schedule: | a) Eligibility according to inclusion and exclusion criteria b) Obtaining signed Informed Consent Form (ICF) c) Demographics (sex, year of birth, smoking status) d) Risk factors & medical history e) Concomitant medications f) Disease oriented physical examination including vital signs (weight, height, BMI, heart rate, blood pressure) and ABI (except in cases |



Document No. CL-003 Version 2.2 

where blood pressure cuff occlusion of the extremity is contraindicated)

- g) Blood test including: RBC, Hemoglobin, WBC, Platelet count, PT, aPTT, INR, serum creatine-kinase isoform MB (CK-MB) and serum creatinine
- h) Pregnancy test, if applicable
- i) Safety evaluation (AE/SAE evaluation)

#### Intervention (Use of WIRION™):

- a) Investigational procedure & materials (atherectomy device, EPS, guide wires and contrast medium)
- b) Intervention details (investigator name, procedure duration and fluoroscopy time)
- c) Angiography of target lesion
- d) Dilation after atherectomy
- e) Stent placement after atherectomy
- f) Angiographic assessment of visible distal embolization, as evidenced by new angiographic filling defect, slow flow, and/or loss of distal tibial runoff
- g) AE/SAE
- h) Usability questionnaire
- i) Visual assessment of debris in the filter
- j) Concomitant medications

#### Pre-Discharge Follow-up:

- a) Disease oriented physical exam including vital signs (heart rate and blood pressure) and ABI (except in cases where blood pressure cuff occlusion of the extremity is contraindicated)
- b) AE/SAE evaluation
- c) Blood test including: RBC, Hemoglobin, WBC, Platelet count, PT, aPTT, INR and serum creatine-kinase isoform MB (CK-MB) and serum creatinine
- d) Concomitant medications

#### **End-of-Study Follow-up Visit** (30±7 days post procedure):

- a) AE/SAE evaluation
- b) Disease oriented physical exam including vital signs (heart rate and blood pressure) and ABI (except in cases where blood pressure cuff occlusion of the extremity is contraindicated)

## Statistical Considerations:

A performance goal group sequential design with a maximum of two stages with rejection boundaries according to Lan-DeMets alpha spending function with O'Brien- Fleming boundaries. The expected proportion of subjects who would meet the primary endpoint if treated according to current clinical practice is 10.7%. This performance goal is based on the DEFINITVE LE and DEFINITVE Ca++ trials.

The study is designed to test the primary null hypothesis that the 30-day MAE outcome using the WIRION<sup>TM</sup> EPS in conjunction with atherectomy is equal to or higher than the PG of 19.26%, as opposed to the alternative hypothesis that the MAE is less than this PG. An interim analysis will be carried out when



Document No. CL-003 Version 2.2 

100 (68.5%) of the originally planned subjects have reached the 30-day follow-up. Using an Exact Binomial Test and under the following assumptions:

Alpha (one-sided) = 0.025  $\beta$ = 0.20PE= 10.7%Performance goal= 19.26%

An estimated 145 evaluable subjects will be required for 80% power if the study reaches the final analysis. With an anticipated combined loss-to-follow-up of up to 5%, 153 patients will be enrolled in the study.

An interim analysis will be performed when 100 subjects (approximately 68.5% of the 145 evaluable subjects) have completed the study; two potential options will be pursued:

The study will be stopped for efficacy if the primary null hypothesis is rejected at one sided alpha = 0.0068 based on the Lan-DeMets alpha spending function with O'Brien - Fleming boundaries.

If based on the interim analysis the primary null hypothesis cannot be rejected, then the trial will continue to a total sample size of 153 enrolled subjects (i.e., 145 evaluable subjects). This test will be conducted at one-sided alpha = 0.0229, in order to control the overall Type I error at 2.5%.

Study success is defined as rejecting the null hypothesis.

**Duration of Study** 

The estimated study duration is ten months, including a recruitment phase and follow up period of 30±7 days